CLINICAL TRIAL: NCT03378622
Title: The Use of Anchor Versus Suturing for Attachment of Vaginal Mesh in Minimally Invasive Sacrocolpopexy
Brief Title: Anchor for Robotic Sacrocolpopexy
Acronym: ARiSe
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11460
Record Dates: First submitted 2017-12-04; First posted 2017-12-20 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anchor (Experimental): Anchor used for mesh attachment
  Interventions: Other: Anchor
- Suture (Active Comparator): Suture used for mesh attachment
  Interventions: Other: Suture

INTERVENTIONS:
Other: Anchor — Anchor technique for mesh attachment
  Arms: Anchor
Other: Suture — Suture technique for mesh attachment
  Arms: Suture

SUMMARY:
1. PRIMARY OBJECTIVE: To assess the effect of absorbable anchor compared to suturing for mesh attachment to vagina in robotic assisted sacrocolpopexy on the length of surgery for this portion of the procedure.
2. SECONDARY OBJECTIVES:

   i. To assess intraoperative and ii. postoperative complication rates, iii. Intraoperative 10 cm visual analog scale (VAS), to subjectively assess surgeon satisfaction with the technique iv. post-operative Pelvic Organ Prolapse Quantification (POPQ) evaluation for anatomic failure and v. a VAS of the vaginal walls overall appearance

DETAILED DESCRIPTION:
By applying a commonly used surgical technique of absorbable anchors to a new surgery, Sacrocolpopexy (SCP), operative time may be decreased while providing similar patient outcomes. Absorbable anchors have been validated in mesh fixation during laparoscopic surgical repair of hernias. This technique potentially takes less time than traditional suturing, thus decreasing cost and morbidity of anesthesia. The investigators hypothesis proposes that for women undergoing SCP at a large managed care organization, participants receiving anchor suture staples to attach the mesh to the vagina compared to participants receiving standard treatment will require 50% shorter surgical time for the mesh attachment portion of the surgery. The investigators secondary hypothesis is for women undergoing SCP at a large managed care organization, participants receiving anchor suture staples to attach the mesh to the vagina compared to participants receiving standard treatment will have similar rates of intra-operative and post-operative complications and surgical failure. On VAS, patients will not have different appearance of the vaginal walls. Surgeons will report higher satisfaction with the anchor technique.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Diagnosis of POP, defined as the descent of one or more of four different anatomic structures, a)the uterus(cervix), b)the apex of the vagina (in those status post hysterectomy) c) the anterior vaginal wall, or d) the posterior vaginal wall. This is defined on exam as the POPQ points Ba, C, or Bp >0 cm beyond the hymen, uterine(cervix) descent into at least the lower half the vagina (defined as point c> -tvl/2) or post hysterectomy vault into the lower 2/3 of the vagina. Bothersome bulge symptoms as indicated on question 3 of the Pelvic Floor Disorder Inventory (PFDI-20) form relating to 'sensation of bulging' or something 'falling out'
* Desire surgical treatment for POP with SCP
* Available for up to 6 months of follow up
* Not pregnant or desiring future pregnancy
* Written informed consent is obtained.

Exclusion Criteria:

* Known adverse reaction to synthetic mesh, or complications including but not limited to erosion, fistula, or abscess.
* Cervical intraepithelial neoplasia (cervical intraepithelial neoplasia (CIN) 2, CIN3, or cancer)
* Unresolved chronic pelvic pain
* Prior abdominal or pelvic radiation
* Contraindications to the surgical procedures including known horseshoe kidney, pelvic abscess or active diverticular abscess or diverticulitis

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 53 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Mesh Attachment Time | Assessed at one time point, during the participants surgery.
  Mesh Attachment Time

SECONDARY OUTCOMES:
Perioperative Complications | Assessed at one time point, during the participants surgery.
  Perioperative Complications
Postoperative Complications | Assessed at two time points, 6 weeks and 6 months postoperatively
  Postoperative Complications
Surgeon Satisfaction | Assessed at one time point, during the participants surgery.
  Surgeon Satisfaction assessed using a visual analog scale (10 point)assessment of satisfaction
Surgical Failure | Assessed at two time points, 6 weeks and 6 months postoperatively
  Surgical Failure assessed using the pelvic organ prolapse quantification scoring system.
Vaginal wall appearance | Assessed at two time points, 6 weeks and 6 months postoperatively
  Vaginal wall appearance assessed using a using a visual analog scale (10 point)assessment of overall appearance as well as sub-categories of anterior and posterior walls.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A Berger, Study Director — Kaiser Permanente; Shawn A Menefee, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanent San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger AA, Tan-Kim J, Menefee SA. Anchor vs suture for the attachment of vaginal mesh in a robotic-assisted sacrocolpopexy: a randomized clinical trial. Am J Obstet Gynecol. 2020 Aug;223(2):258.e1-258.e8. doi: 10.1016/j.ajog.2020.05.018. Epub 2020 May 13. PMID 32413431

DOCUMENTS (3):
  • Informed Consent Form (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03378622/ICF_000.pdf
  • Study Protocol (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03378622/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03378622/SAP_002.pdf